CLINICAL TRIAL: NCT00056979
Title: Anti-CD45 (YTH-24 & YTH 54) and ANTI-CD52 (CAMPATH-1H) Monoclonal Antibody Conditioning Regimen for Allogeneic Stem Cell Transplantation of Patients With Inherited Metabolic Storage Diseases
Brief Title: Monoclonal Antibody Conditioning for Allogeneic Stem Cell Transplantation of Patients With Inherited Metabolic Storage Diseases
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Robert Krance, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H11909; MAID
Record Dates: First submitted 2003-03-26; First posted 2003-03-27 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Inherited Metabolic Storage Diseases
Keywords: Metabolic diseases
MeSH Terms: conditions — Metabolic Diseases | interventions — Alemtuzumab; Tacrolimus; fludarabine

ARMS (1):
- Fludarabine, CAMPATH-1H , Anti-CD45, FK506 (Experimental): Fludarabine will be given as a daily IV (intravenous, by vein) infusion for a total of 5 days. CAMPATH-1H will be given as a daily 4-hour IV (intravenous, by vein) infusion for three days. Anti-CD45 will be given as a daily 6-hour IV infusion over the next 4 days. To help prevent body from rejecting the transplant, the drug FK506 will be given, starting two days before the transplant and continuing for three months.
  Interventions: Drug: CAMPATH-1H; Drug: Anti-CD45; Drug: FK506; Drug: Fludarabine

INTERVENTIONS:
Drug: CAMPATH-1H
Drug: Anti-CD45
Drug: FK506
Drug: Fludarabine

SUMMARY:
This study treats patients with an inherited disease that prevents the body from making a specific protein or enzyme needed for the body's metabolism. Lack of this enzyme causes accumulation of harmful or toxic substances in the body, which leads to deterioration and failure of organs such as the brain or the heart. This disease can be fatal.

Some patients with inherited metabolic storage disease may benefit from an allogeneic stem cell transplant ('allogeneic' means that the stem cells come from another person). Stem cells are created in the bone marrow. They mature into different types of blood cells that are needed including red blood cells, white blood cells, and platelets. Stem cells, when transplanted, can make a new blood system. Donor stem cells can make the protein or enzyme patients with this disease cells cannot. The donor cells may prevent further accumulation of toxic substances. It is hoped that the donor cells can prevent or stop the disease from progressing.

This research study uses a new pre-treatment combination of two drugs, Anti-CD45 and CAMPATH-1H. Anti-CD45 and CAMPATH-1H are antibodies against certain types of blood cells. CAMPATH-1H is particularly important because it stays active in the body for a long time after infusion, which means it may work longer at preventing GVHD symptoms. In addition to antibodies, patients will receive Fludarabine, which is a chemotherapy drug. Fludarabine kills bone marrow cells and is given to reduce the bone marrow cells so that donor stem cells may 'take.'

DETAILED DESCRIPTION:
Fludarabine will be given as a daily IV (intravenous, by vein) infusion for a total of 5 days. CAMPATH-1H will be given as a daily 4-hour IV (intravenous, by vein) infusion for three days. Anti-CD45 will be given as a daily 6-hour IV infusion over the next 4 days. Then patients will have a one-day rest period before receiving the stem cell transplant. To help prevent the body from rejecting the transplant, patients will also receive the drug FK506, starting two days before the transplant and continuing for three months. If there is no GVHD, the amount of FK506 patients are taking will be reduced by 20% every 2 weeks until this medication is stopped.

ELIGIBILITY:
Inclusion criteria:

* Patients with inherited metabolic storage diseases of all ages are eligible.
* Diagnosis of inherited metabolic storage disease confirmed by standard biochemical and genetic studies in consultation with the Department of Genetics at the Baylor College of Medicine
* Inherited metabolic storage diseases which may be stabilized or improved by stem cell transplantation include: Hurler, Hunter, Maroteaux-Lamy, Sly, Wolman, Gaucher, Farber, Nieman-Pick, Mannosidosis, Aspartylglucosaminuria, Fucosidosis, Neuronal Ceroid-Lipofuscinosis, Metachromatic Leukodystrophy, Globoid Cell Leukodystrophy, and Adrenoleukodystrophy
* Availability of an HLA matched or mismatched (up to one haplotype) donor who is not an obligate carrier for the inherited condition or an unrelated HLA matched stem cell donor. Fully matched is defined as 6/6 match by high resolution DR based DNA typing.
* Female patients of childbearing age must have a negative pregnancy test and be willing to use an effective means of birth control.

Exclusion criteria:

* Patients with a life expectancy (<6 weeks) limited by diseases other than inherited metabolic storage disease
* Patients with advanced inherited metabolic storage disease, which has not been stabilized or improved by hematopoietic stem cell transplantation.
* Patients with symptomatic cardiac disease, or evidence of significant cardiac disease by echocardiogram (i.e., shortening fraction <25%)
* Patients with severe renal disease (Creatinine >2 x normal for age)
* Patients with known allergy to rat serum products
* Patients with a Karnofsky or Lansky score <50%.
* Patients with a severe infection that on evaluation by the Principal Investigator precludes ablative chemotherapy or successful transplantation
* Patients with severe personality disorder or mental illness or neuropsychological evaluation indicating too much damage for the transplant to be of benefit.
* Patients with documented HIV positivity.
* Patients with grade III-IV liver toxicity not related to metabolic storage disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2002-06; Primary Completion 2003-06 (Actual); Study Completion 2003-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm K Brenner, MD, Study Chair — Baylor College of Medicine
Locations (2):
- United States (2):
  - Texas Children's Hospital, Houston, Texas
  - The Methodist Hospital, Houston, Texas